CLINICAL TRIAL: NCT04327544
Title: Nutritional Education and Exercise Intervention in Preventing Frailty Among Pre-frail Malaysian Elderly in PPR Flats Kuala Lumpur
Brief Title: A Health Promotion Program to Prevent Frailty and Improve Frailty Status Among Pre-frail Elderly: Frailty Intervention Through Nutrition Education and Exercises.
Acronym: FINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Nurul Izzati binti Mohd Suffian, Principle Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GP-IPS/2017/9547700
Record Dates: First submitted 2020-02-23; First posted 2020-03-31 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Frail Elderly Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frailty Intervention group (Experimental): A multi-domain intervention program that includes nutrition education and low to moderate multi-component exercise intervention.
  Interventions: Behavioral: Frailty Intervention
- Control group (No Intervention): Respondents in the control group will not receive any nutritional education or exercise intervention activities.

INTERVENTIONS:
Behavioral: Frailty Intervention — In overall, participants will attend one session of frailty talk, 22 sessions of low to moderate intensity of multi-components exercise course and 6 session of nutrition education interventions. Both nutritional education and exercise intervention will be conducted concurrently for a 12-week (3-month) of intervention period. Noted that every session will be held in PPR flats' facility area or hall around 60 minutes that will be conducted by the dietitian or nutritionist and physiotherapist from the research team.
  Other Names: FITNESS
  Arms: Frailty Intervention group

SUMMARY:
Prevention of frailty is a major concern in geriatrics due to its high prevalence and various adverse health outcomes among elderly population. This two phases of study aims to develop, implement and evaluate the effectiveness of nutritional education and exercise intervention among pre-frail Malaysian elderly. In the first phase of the study, the frailty intervention module and educational materials (flipchart, PowerPoint slides, booklet and posters) for the frailty intervention program will be developed based on extensive literature review and discussions with research group (dietitians, nutritionists, physiotherapists and medical doctor). The module will be developed to provide knowledge and skills to health practitioners in order to conduct the program towards pre-frail elderly, while the educational materials will aid health practitioners and the elderlies in teaching and learning process respectively. Evaluation for acceptability of frailty intervention module and educational materials will also be conducted in phase 1 study. The second phase of the study will be a three- month (12 weeks), single-blind, two-armed, cluster randomised controlled trial (cluster RCT) research to evaluate the effects of combined nutritional education and exercise intervention among pre-frail elderly in PPR flats Kuala Lumpur. Screening of the pre-frail status among the elderly in PPR flats Kuala Lumpur will be conducted in order to recruit subjects who match the inclusion criteria to join the intervention program. Evaluation will be performed during pre-intervention (1 week before intervention starts), post-intervention (3 month immediate after intervention starts) and 3-month follow-up (3 months after post-intervention). The frailty intervention includes both nutritional education and low-intensity exercise intervention. Generally, respondents in the intervention group will received the developed educational materials and participate in healthy eating talk, group diet counselling, multicomponent exercise sessions. In short, the interventions being examined will provide major potential benefits to the older population in terms of preventing transition to frailty and potentially reduce adverse health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Man or women aged 60 years and above
* Meet one or two frailty phenotype score (pre-frail)
* Able to ambulate without personal assistance
* Residing in the PPR flats in Kuala Lumpur
* Willing to participate in the intervention program with informed consent

Exclusion Criteria:

* Self-reported chronic diseases (heart-related disease, COPD, stroke, cancer, asthma, renal dysfunction, terminally ill)
* PAR-Q & YOU questionnaire (Yes≥1)
* Bedridden
* Cognitive impairment (ECAQ<6)
* Sensory impairment (visual & hearing) that will interfere with communication
* Unable to read and write
* Already involved or still participating in any health interventional studies
* Any sustained fracture (hip, vertebrata) in past six month
* Any surgery (hip, abdominal area) in past six months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Changes in Frailty score | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  Frailty score will be assessed using the well-established Malay language standardized phenotype of frailty questionnaire as proposed by Fried et al. The questionnaire evaluates five components of the frailty syndrome (weight loss, exhaustion, weakness, slowness and low activity) and allocates one point for each criterion met. The highest the score indicate worst condition of the elderly in term of frailty.
Changes of Frailty status | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  Frailty status will be assessed using the well-established Malay language standardised phenotype of frailty questionnaire as proposed by Fried et al. The questionnaire evaluates five components of the frailty syndrome (weight loss, exhaustion, weakness, slowness and low activity) and allocates one point for each criterion met; respondents meeting zero criteria are defined as non-frail (normal), whereas those meeting one or two criteria are defined as pre-frail, and those meeting three, four or five criteria are defined as frail

SECONDARY OUTCOMES:
Changes in knowledge, attitude and practice (KAP) towards frailty, nutrition and exercise | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  The KAP questions will be developed prior to data collection to measure the construct of knowledge, attitude and practice in relation to frailty, nutrition and exercise among elderly. The questions consisted of items based on the content of the developed educational materials. A validation and reliability study will be conducted after it is developed. The result will be in term of score. The higher score in knowledge indicate better knowledge. Higher score in attitude indicate more positive attitude and higher score in practice indicate healthier lifestyle practice by the participant.
Changes in dietary intake | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  The amount of food items consumed by the respondents in the past week will be recorded by the validated Malay language of Diet History Questionnaire (DHQ) via interview method. The data will be analysed using the Nutritionist Pro TM Diet Analysis Software, then will be compared to the Malaysian Recommended Nutrient intake.
Changes in cognitive status | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  This study will used the validated Malay language version of Mini-Mental State Examination (M-MMSE) questionnaire to assess the cognitive functioning of the respondents. The M-MMSE is an 11-question measure that tests five areas of cognitive function: orientation (2 items), registration (1 item), attention and calculation (1 item), recall (1 item), and language (6 items). The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment.
Changes in functional ability | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  The well-established Malay language of Lawton Instrumental Activities of Daily Living (IADL) questionnaire will be used to assess the respondents' ability to perform eight daily activities (i.e. ability to use telephone, shopping, preparing meals, housekeeping, doing laundry, using public transport, taking medications, and handling finances). Presence of 'functional disability' will be defined as having difficulty or needing help in at least one of these 8 items IADL activities, while normal functioning will be defined if one can perform all 8 activities independently.
Changes in mobility status | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  A well-established Malay language of Short Physical Performance Battery (SPPB) will be used for this study to test the respondents' mobility status to evaluate lower limb extremity functioning in three components (balance test, gait speed test and repeated chair stand test). There are three components namely: 1) balance test (the ability to stand for 10 sec with the feet together in the side-by-side, semi-tandem, and tandem positions) 2) gait speed test (time to walk 4 metres) and 3) repeated chair stand test (time to rise from a chair and return to the seated position 5 times). A score ranging from 0 to 4 (0=inability to complete the task; 4=highest level of function) will be scored for each task of SPPB with the sum of these three tests (0-12) reflecting the complete measurement of physical function. Thus, lower scores on the SPPB reflect higher odds of mobility-related disability.
Changes in risk of falls | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  The Malay language of Berg Balance Scale (BBS) will be used to assess the risk of falls among the respondents by assessing the performance of 14 different functional tasks. The different tasks including ability to sit, stand, reach, lean over, turn and look over each shoulder, turn in a complete circle, and step. The BBS, which rates each performance from 0 (cannot perform) to 4 (normal performance), with the total possible score on the BBS is 56, indicating excellent balance. The presence of high risk of falls will be scored within 0-20.
Changes in body mass index | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  Body Mass Index (BMI) will be calculated as weight (kg) divided by the square of the height (m2) of either standing height or alternative height. The classification for BMI is based on World Health Organization; value of less than 18.5 kg/m2 and more than 24.9 kg/m2 indicates underweight and overweight respectively. Seca 803 Digital Weight Scale will be used to measure body weight of the respondents in light clothing (without shoes) to the nearest 0.1 kilogram. Standing height will be taken using SECA portable stadiometer (SECA-213 model) to the nearest 0.1 centimeter with the subject standing barefoot. Subjects who are found to have kyphosis problem or difficulty to stand straight will be replaced with alternative height (demi-span) measurement using equations developed among Malaysian elderly.
Changes in mid upper arm circumference (MUAC) | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  Body part circumference, MUAC will be measured using a flexible non-stretchable tape (SECA-201 model). MUAC is measured to indicate the loss of peripheral muscle mass and is an indicator for upper-body muscle mass and recommended to use to assess the nutritional status of elderly. MUAC need to identify the midpoint of the bare non-dominant arm first, then measure circumference comfortably round the arm at the midpoint. Reading will be taken twice to the nearest 0.1cm and average circumference will be calculated. A MUAC value of less than 23.0 cm for men and 22.0 cm for women indicates loss of peripheral muscle mass.
Changes in calf circumference (CC) | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  Body part circumference, CC will be measured using a flexible non-stretchable tape (SECA-201 model). CC measurement is to indicate muscle loss especially in the lower limb and considered a pertinent marker of the nutritional status in the elderly. For CC, the measuring tape will be wrapped comfortably around the calf (non-dominant leg) at the widest part while respondents are sitting down and recorded to the nearest 0.1cm. The criterion to indicate muscle loss, especially in the lower limb was based on the local classification for Malaysian elderly with a value of less than 30.1 cm for men and 27.3 cm for women respectively.
Changes in percentage of total body fat (%TBF) | The measurement will be conducted three times; pre- intervention (1 week before intervention start), post - intervention (immediately after intervention end) and at 3 months follow - up (3 months after post intervention).
  The %TBF refers to the amount of body fat mass in regard to the total body weight expressed as a percentage. It will be determined by the OMRON body fat analyzer (HBF-375 model). Prior to the measurement, respondents will be ensured to remove all metal accessories (i.e. necklace, rings, earrings, watch, cell phones and bracelets) that might interfere the reading. Information like age, gender and height will be set into the analyzer. Respondents will be required to stand on weighing platform with bare feet in contact with the metal parts while both hands holding tightly the grip electrodes with outstretched arms. The %TBF of the respondents will be classified into certain ranges for person 18 years of age and older. %TBF that is low than 5 and 8 indicate too low muscle while more than 25 and 32 indicate too high for male and female respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Siti Nur'Asyura binti Adznam, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Projek Perumahan Rakyat (PPR), Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No